CLINICAL TRIAL: NCT01374659
Title: Effectiveness of [124I]-PET/CT and [18F]-FDG-PET/CT for Localizing Recurrence in Patients With Differentiated Thyroid Carcinoma Who Have Elevated Serum Thyroglobulin Levels But Are Tumor-negative on Conventional Imaging Studies
Brief Title: Diagnostic Utility of [18F]-FDG-PET/CT and [124I]-PET/CT for Detection of Recurrence in Differentiated Thyroid Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Korean Association of Endocrine Surgeons (Network)
Responsible Party: Ajou University Medical Center, Department of Surgery, Korean Association of Endocrine Surgeons
Other Study IDs: Korean AES007
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-01

CONDITIONS: Thyroid Cancer; Recurrence
Keywords: 124-I PET; FDG-PET; PET/CT; recurrence; differentiated thyroid carcinoma; diagnostic value
MeSH Terms: conditions — Thyroid Neoplasms; Recurrence

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Study patients: Study patients with histologically proven DTC were studied. All patients had previously undergone total thyroidectomy and more than one session of postoperative RI therapy. After the last RI therapy session, all patients showed increasing pathological Tg levels (Tg > 9-10 ng/ml) after TSH stimulation (TSH > 30 mU/l). However, neither tumor recurrence nor metastasis could be detected in any patient by post-therapeutic [131I] scanning, neck US, or chest radiography. Patients with obvious cervical pathology or positive fine-needle aspiration cytology (FNAC) were excluded from the study. The work was approved by our Institutional Review Board and written informed consent was obtained from each patient.

SUMMARY:
Several studies have indicated that [124I]-PET/CT or [18F]-FDG-PET/CT may be useful to locate recurrent differentiated thyroid carcinoma lesions in patients with elevated thyroglobulin levels but who do not show pathological lesions when conventional imaging modalities are used. Thus, the investigators evaluated the effectiveness of PET/CT using both [124I] and [18F]-FDG in such patients.

DETAILED DESCRIPTION:
<Inclusion Criteria> Patients with histologically proven DTC were studied. All patients had previously undergone total thyroidectomy and more than one session of postoperative RI therapy. More than 12 months of follow-up after the last RI therapy session, all patients showed increasing pathological Tg levels (Tg > 9-10 ng/ml) after TSH stimulation (TSH > 30 mU/l). However, neither tumor recurrence nor metastasis could be detected in any patient by post-therapeutic [131I] scanning, neck US, or chest radiography. Patients with obvious cervical pathology or positive fine-needle aspiration cytology (FNAC) were excluded from the study. The work was approved by our Institutional Review Board and written informed consent was obtained from each patient.

<Study protocol> The study was prospectively designed to evaluate the diagnostic efficacies of [18F]-FDG-PET/CT and [124I]-PET/CT in patients with elevated Tg levels, but who yielded no pathological findings on conventional imaging. The [124I] radioisotope was supplied by the Radiopharmaceutical Research Team of the Korea Institute of Radiological and Medical Sciences (KIRAMS). All involved patients underwent a diagnostic [131I] scan, [18F]-FDG-PET/CT, and [124I]-PET/CT. On the first day (D1) of the study, blood and urine were collected for routine examination; to measure blood TSH, Tg, and anti-Tg antibody levels; and to assess urine iodine excretion after 4 weeks of levothyroxine (LT4) withdrawal. All patients had consumed a low-iodine diet for the prior 2 weeks, following written instructions and assisted by a dietician. On the second day (D2) of the study, an [131I] scan was obtained 48 h after administration of 74 MBq of [131I]. On day 10 (D10) of the study, patients fasted for at least 4 h before examination, and were (intravenously) given 370 MBq [18F]-FDG. All patients were instructed to rest comfortably for 60 min and to empty the bladder before scanning. Whole-body PET/CT images were obtained using a Discovery ST scanner (GE Healthcare, Milwaukee, WI). Seven or eight frames (3 min/frame) of emission PET data were acquired in the two-dimensional mode after noncontrast CT scans had been performed from the base of the skull to the upper thigh (tube rotation time of 1 s per revolution; 120 kV; 60 mA; 7.5 mm per rotation; and an acquisition time of 60.9 s for a scan length of 867 mm). Emission PET images were reconstructed via non-contrast CT using an iterative method (ordered-subsets expectation maximization with two iterations and 30 subsets; field of view 600 mm; slice thickness 3.27 mm). Attenuation-corrected PET/CT images were reviewed on an Xeleris workstation (GE Healthcare). All images were independently interpreted by two experienced nuclear medicine physicians and screened for "hot spots" indicative of hypermetabolic abnormalities.

On day 11 (D11) of the study, 24 h after administration of an [124I] trace dose (74 MBq), whole-body PET/CT scans were obtained using the Discovery ST scanner. First, a non-enhanced CT scan was performed, from the base of the skull to the upper thigh (tube rotation time of 1 s per revolution; 140 kV; 80 mA; 3.75 mm per rotation; acquisition time of 23.9 s for a scan length of 804 mm). Subsequently, seven or eight frames (5 min per frame) of emission PET data were acquired in the two-dimensional mode and reconstructed via CT using an iterative method (software from General Electric Medical Systems; ordered-subsets expectation maximization with two iterations and 21 subsets; field of view 600 mm; slice thickness 3.27 mm).

<Data analysis> To ensure that the interpretation of [18F]-FDG-PET/CT and [124I]-PET/CT data was performed under similar conditions, all physicians who initially read images of one type were deliberately blinded to the results of the other type of imaging, and to patient clinical data. This was achieved by ensuring that the interpreting physicians were not involved in patient clinical care. Findings on [18F]-FDG-PET and [124I]-PET scanning were compared with data from diagnostic and post-therapeutic [131I] scans. Moreover, the data were compared with those of radiological imaging (US, CT, and MRI information), and/or those of cytological investigation (FNAC), to confirm (or otherwise) the findings of the [131I] scans, and those of both forms of PET/CT (using [18F]-FDG and [124I]). For each patient, the presence or absence, and number and localization of any recurrent lesions (if present) were determined. The data of both types of PET/CT scans were classified as follows: 1) True-positive, if pathologic [18F]-FDG or [124I] uptake was proven by histology, cytology, or other imaging techniques, and caused therapy to be changed; 2) False-positive, if no pathologic [18F]-FDG or [124I] uptake was seen (such observations were of no clinical consequence); 3) True-negative, if no [18F]-FDG or [124I] uptake was found and the patient had neither an elevated Tg level nor any evidence of recurrence upon subsequent follow-up; and, 4) False-negative if no [18F]-FDG or [124I] uptake was noted despite elevated Tg levels, even if positive findings were obtained when other imaging methods were employed.

ELIGIBILITY:
Inclusion Criteria:

* Study patients with histologically proven DTC were studied. All patients had previously undergone total thyroidectomy and more than one session of postoperative RI therapy.During follow-up after the last RI therapy session, all patients showed increasing pathological Tg levels (Tg > 9-10 ng/ml) after TSH stimulation (TSH > 30 mU/l). However, neither tumor recurrence nor metastasis could be detected in any patient by post-therapeutic [131I] scanning, neck US, or chest radiography.

Exclusion Criteria:

* Patients with obvious cervical pathology or positive fine-needle aspiration cytology (FNAC) were excluded from the study. The work was approved by our Institutional Review Board and written informed consent was obtained from each patient.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study patients who underwent total thyroidectomy with more than one of high dose radioactive iodine treatment, showed elevated Tg levels, but who yielded no pathological findings on conventional imaging during follow-up period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-06 (Actual); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Diagnostic values of [124I]-PET/CT and [18F]-FDG-PET/CT imaging | Follow up in more than 10 months after treatment
  1) True-positive, if pathologic [18F]-FDG or [124I] uptake(;PET-uptake) was proven by histology, cytology, or other imaging techniques, and caused therapy to be changed; 2) False-positive, if no pathologic PET-uptake was seen; 3) True-negative, if no PET-uptake was found and the patient had neither an elevated Tg level nor any evidence of recurrence upon subsequent follow-up; and, 4) False-negative if no PET-uptake was noted despite elevated Tg levels, even if positive findings were obtained when other imaging methods were employed.

CONTACTS AND LOCATIONS:
Overall Officials: Jandee Lee, MD, Principal Investigator — Korean Association of Endocrine Surgeons
Locations (1):
- Jandee Lee, Suwon, South Korea